CLINICAL TRIAL: NCT00548158
Title: Preliminary Safety Study of Pioglitazone Therapy for Diabetes on Macular Thickness and Vision in Type 2 Diabetes
Brief Title: Effect of Pioglitazone Therapy for Type 2 Diabetes on Vision
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Other Study IDs: DUB-071127
Record Dates: First submitted 2007-10-19; First posted 2007-10-23 (Estimated); Last update posted 2007-10-23 (Estimated); Status verified 2007-10

CONDITIONS: Type 2 Diabetes
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We are studying patients with diabetes who under proper medical care and administer an approved drug. Our interest is if this drug has any sideeffect on vision and if this drug may cause swelling of the retina.

DETAILED DESCRIPTION:
To evaluate the safety of pioglitazone treatment for diabetes. Recent reports suggest that oral glitazone treatment may cause or exacerbate retinal edema. We hypothesized that glitazone treatment may cause subclinical edema evidenced by increased retinal thickness. We will conduct a double-masked, prospective safety study of 19 subjects undergoing placebo-controlled treatment with pioglitazone. Patient treatment consisted of either insulin with placebo or insulin with pioglitazone. The main outcome measures are ETDRS visual acuity and retinal thickness measured with optical coherence tomography.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with type 2 diabetes mellitus on insulin therapy, 30-75 years of age with Hgb 1c values between 7.5 - 10% and a BMI of < 40kg/m2.
* Patients were enrolled if they have been on a stable anti-hypertensive and lipid regimen for 90 days prior to study randomization.
* Patients must have had the ability to understand the requirements of the study, provide written consent and agree to abide by study requirements.

Exclusion Criteria:

* Prior treatment with sulfonylurea, or metformin within 21 days before study entry, prior treatment with NSAIDs, or diuretics within 21 days of screening, serum creatinine levels above 1.5 mg/dl for males or above 1.4 for females or creatinine clearance less than 70 ml/min by Cockcroft and Gault, or serum albumin levels of less than 2.5 gm/dl.
* Other exclusion criteria were elevated hepatic enzymes (aspartate aminotransferase or alanine aminotransferase more than 2.5 times upper limit of normal) or uncontrolled or untreated significant pulmonary, neurological condition, or cardiovascular disease, including hypertension, congestive heart failure (specifically New York Heart Association Type III or IV patients), angina, peripheral vascular disease, or greater than +1 peripheral edema.
* Furthermore, any patients with any condition that would jeopardize their safety or affect the validity of the trial results were excluded from this study.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients with type 2 diabetes mellitus on insulin therapy, 30-75 years of age with Hgb 1c values between 7.5 - 10% and a BMI of < 40kg/m2. Patients were enrolled if they have been on a stable anti-hypertensive and lipid regimen for 90 days prior to study randomization.
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2004-10; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
ETDRS visual acuity | baseline and at 3 months followup visit

SECONDARY OUTCOMES:
retinal thickness measured by OCT | baseline and at 3 months followup visit

CONTACTS AND LOCATIONS:
Overall Officials: William R Freeman, MD, Principal Investigator — University of California, San Diego